CLINICAL TRIAL: NCT00749931
Title: MarginProbe, a Device for Intraoperative Assessment of Margin Status in Breast Conservation Surgery
Acronym: Pivotal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dune Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CP-03-001
Record Dates: First submitted 2008-09-07; First posted 2008-09-09 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Breast Cancer
Keywords: IDC, DCIS, ILC
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOC (Active Comparator): Standard of Care arm - standard of care lumpectomy procedure
  Interventions: Procedure: Lumpectomy
- Device + SOC (Experimental): Use of the device in addition to the standard of care lumpectomy procedure.
  Interventions: Device: MarginProbe; Procedure: Lumpectomy

INTERVENTIONS:
Device: MarginProbe — Device use to assess margin status of the excised specimen surface.
  Arms: Device + SOC
Procedure: Lumpectomy — Standard of care lumpectomy procedure

SUMMARY:
The purpose of this study is to show that addition of device use to a routine breast cancer tumor excision procedure is beneficial and assists the surgeon in correctly determining the extent of excision.

DETAILED DESCRIPTION:
The study is a prospective, multi-center, randomized, double arm study demonstrating the effectiveness of the device in adjunctive use for locating the tissue for additional excision following primary specimen excision. One arm is a "Standard of Care" (SOC) Control group and the other arm a "Device+SOC" group.In the "Device +SOC" group the surgeon will use the MarginProbe device on the tissue specimen removed during the surgical procedure.The surgeon will use the results derived from the device and other routine assessments to decide if it is necessary to remove some additional breast tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Women histologically diagnosed with carcinoma of the breast
2. Women with non-palpable malignant lesions, requiring image guided localization.
3. Undergoing lumpectomy (partial mastectomy) procedure.
4. Age 18 years or more
5. Signed ICF

Exclusion Criteria:

1. Multicentric disease (histologically diagnosed cancer in two different quadrants of the breast)
2. Bilateral disease (diagnosed cancer in both breasts)
3. Neoadjuvant systemic therapy
4. Previous radiation in the operated breast
5. Prior surgical procedure in the same breast
6. Implants in the operated breast
7. Pregnancy
8. Lactation
9. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanir M. Allweis, MD, Principal Investigator — Hadassah Medical Organization, Israel; Moshe Carmon, MD, Principal Investigator — Shaare Zedek Medical Center, Israel; Tami Karni, MD, Principal Investigator — Assaf Harefeh Medical Center, Israel; Alison Estabrook, MD, Principal Investigator — St. Luke's Roosevelt, NY, USA; Freya Schnabel, MD, Principal Investigator — NYU Clinical Cancer Center, NY, USA; Rache M. Simmons, MD, Principal Investigator — Weill Medical College of Cornell University, NY, USA; Sheldon M. Feldman, MD, Principal Investigator — Columbia University Medical Center, NY, USA; Mark A. Gittelman, MD, Principal Investigator — Breast Care Specialist, Allentown, Pennsylvania, USA; Neil Friedman, MD, Principal Investigator — Mercy Health Srvices, Baltimore, USA; Kristen L. Fernandez, MD, Principal Investigator — Franklin Square Hospital Center, Baltimore, USA; Shawna C. Willey, MD, Principal Investigator — Georgetown University Hospital, Washington, USA; Lorraine Tafra, MD, Principal Investigator — Anne Arundel Medical Center, Annapolis, USA; Karen Lane, MD, Principal Investigator — UCIrvine Medical Center, California, USA; Jay Harness, MD, Principal Investigator — St. Joseph Hospital, California, USA; Alice Police, MD, Principal Investigator — Pacific Breast Care, California, USA; Dennis R. Holmes, MD, Principal Investigator — University of South California, California, USA; Scott Karlan, MD, Principal Investigator — Cedars Sinai Hospital, California, USA; Stephanie Akbari, MD, Principal Investigator — Virginia Hospital Center; Thomas Frazier, MD, Principal Investigator — Bryn Mawr Hospital; Lisa E. Guerra, MD, Principal Investigator — HOAG Memorial Hospital; Susan K. Boolbol, MD, Principal Investigator — Beth Israel Medical Center, NY, USA
Locations (21):
- United States (18):
  - Pacific Breast Care, Costa Mesa, California
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Hospital, Los Angeles, California
  - HOAG Memorial Hospital, Newport Beach, California
  - St. Joseph Hospital, Orange, California
  - UCIrvine Medical Center, Orange, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Mercy Hospital Services, Baltimore, Maryland
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Beth Israel Medical Center, New York, New York
  - NYU Clinical Cancer Center, New York, New York
  - St. Luke's Roosevelt, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Columbia University Medical Center, New York, New York
  - Breast Care Center, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Virginia Hospital Center, Arlington, Virginia
- Israel (3):
  - Haddasah Medical Organization, Jerusalem
  - Shaare Zedek, Jerusalem
  - Assaf Harofeh Medical Center, Zrifin

REFERENCES:
- [Result] Schnabel F, Boolbol SK, Gittleman M, Karni T, Tafra L, Feldman S, Police A, Friedman NB, Karlan S, Holmes D, Willey SC, Carmon M, Fernandez K, Akbari S, Harness J, Guerra L, Frazier T, Lane K, Simmons RM, Estabrook A, Allweis T. A randomized prospective study of lumpectomy margin assessment with use of MarginProbe in patients with nonpalpable breast malignancies. Ann Surg Oncol. 2014 May;21(5):1589-95. doi: 10.1245/s10434-014-3602-0. Epub 2014 Mar 5. PMID 24595800
- See also: Dune Medical Devices official web site — http://www.dunemedical.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care (SOC): Standard of Care arm - standard of care lumpectomy procedure
  Lumpectomy: Standard of care lumpectomy procedure
- Device + (Standard of Care) SOC; Roll-in: Use of the device in addition to the standard of care lumpectomy procedure.
  MarginProbe: Device use to assess margin status of the excised specimen surface.
  Lumpectomy: Standard of care lumpectomy procedure
Period: Overall Study
Arm/Group | Standard of Care (SOC) | Device + (Standard of Care) SOC | Roll-in
Started | 298 | 298 | 68
Completed | 298 | 298 | 68
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | Device + (Standard of Care) SOC | Total
Number analyzed (Participants) | 298 | 298 | 596
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (11.1) | 60.3 (11.4) | 60.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 298 | 298 | 596
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Effectiveness Endpoint is a Measure of Intraoperative Success in Addressing Positive Margins as Detected by Permanent Pathology)by Additional Oriented Tissue Re-excision From the Surgical Cavity.
Description: Tests the efficacy of the device to intra-operatively assess positive margins (superiority) - CSR is 'positive' when all positive margins, as detected by histology, on the main specimen addressed intra-operatively
Time Frame: two weeks after surgery
Population: The Analysis Set for evaluating intraoperative assessment consisted of patients with at least one histologically positive margin on main lumpectomy specimen ("PSS" - Positive specimen subjects)
Measure: Number; unit: percentage of participants analyzed
Arm/Group | Standard of Care (SOC) | Device + (Standard of Care) SOC
Number analyzed (Participants) | 147 | 163
percentage of participants analyzed | 22.4 | 71.8
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs Device + (Standard of Care) SOC; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Post Hoc Outcome: Re-excision Lumpectomy Procedures Due to Positive Margin on Main Specimens
Time Frame: Up to 2 months post-surgery
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care (SOC) | Device + (Standard of Care) SOC
Number analyzed (Participants) | 298 | 298
percentage of participants | 20.8 | 10.0
Statistical Analysis 1: Comparison: Standard of Care (SOC) vs Device + (Standard of Care) SOC; Test type: Superiority or Other; p = 0.002, Fisher Exact; Relative reduction = .47

ADVERSE EVENTS:
Time Frame: Up to 2 months post-surgery.
Arm/Group | Standard of Care (SOC) | Device + (Standard of Care) SOC | Roll-in
Serious Adverse Events (participants affected / at risk) | 5/298 | 6/298 | 3/68
Other Adverse Events (participants affected / at risk) | 0/298 | 0/298 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=298) | Device + (Standard of Care) SOC (N=298) | Roll-in (N=68)
Infections and infestations (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No